CLINICAL TRIAL: NCT03432741
Title: Pilot Safety and Feasibility Study of an In Vivo Sensitivity Screen Using a Direct Tumor Microinjection Technique and FDG-PET
Brief Title: Direct Tumor Microinjection and FDG-PET in Testing Drug Sensitivity in Patients With Relapsed or Refractory Non-Hodgkin Lymphoma, Hodgkin Lymphoma, or Stage IV Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: funding - sponsor filing Chapter 11 bankruptcy
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1689; NCI-2018-00149 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1689 (Other: Mayo Clinic in Rochester); 16-009337 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2018-02-08; First posted 2018-02-14 (Actual); Last update posted 2025-05-26 (Actual); Status verified 2025-05

CONDITIONS: Breast Adenocarcinoma; Metastatic Breast Carcinoma; Recurrent Breast Carcinoma; Recurrent Hodgkin Lymphoma; Recurrent Mycosis Fungoides; Recurrent Non-Hodgkin Lymphoma; Recurrent Primary Cutaneous T-Cell Non-Hodgkin Lymphoma; Refractory Breast Carcinoma; Refractory Hodgkin Lymphoma; Refractory Mycosis Fungoides; Refractory Nodal Marginal Zone Lymphoma; Refractory Non-Hodgkin Lymphoma; Refractory Primary Cutaneous T-Cell Non-Hodgkin Lymphoma; Stage IV Breast Cancer AJCC v6 and v7
MeSH Terms: conditions — Breast Neoplasms; Hodgkin Disease; Mycosis Fungoides; Lymphoma, Non-Hodgkin; Lymphoma, T-Cell, Cutaneous; Lymphoma, B-Cell, Marginal Zone | interventions — belinostat; carfilzomib; copanlisib; daratumumab; Fluorodeoxyglucose F18; Gemcitabine; Nivolumab; obinutuzumab; pembrolizumab; Magnetic Resonance Spectroscopy; Rituximab; CT-P10; romidepsin; Depsipeptides; Lactones; Sodium Chloride; Trastuzumab; PF-05280014; Ogivri; Ontruzant; trastuzumab biosimilar HLX02

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (FDG-PET, direct tumor microinjection) (Experimental): Patients undergo FDG-PET and receive saline intralesionally on day 1. Patients also receive up to five additional injections of gemcitabine hydrochloride, romidepsin, belinostat, carfilzomib, copanlisib hydrochloride, nivolumab, trastuzumab, daratumumab, obinutuzumab, pembrolizumab, or rituximab intralesionally per investigator on day 1. Beginning 5 days later, patients with nodal/extranodal mass undergo restaging FDG-PET and biopsy (if clinically feasible). Within 3-7 days, patients with cutaneous disease undergo restaging photography and biopsy.
  Interventions: Drug: Belinostat; Drug: Carfilzomib; Drug: Copanlisib Hydrochloride; Biological: Daratumumab; Drug: Fludeoxyglucose F-18; Drug: Gemcitabine Hydrochloride; Other: Laboratory Biomarker Analysis; Biological: Nivolumab; Biological: Obinutuzumab; Biological: Pembrolizumab; Procedure: Positron Emission Tomography; Biological: Rituximab; Drug: Romidepsin; Other: Saline; Biological: Trastuzumab

INTERVENTIONS:
Drug: Belinostat — Given intralesionally
  Other Names: Beleodaq; PXD 101; PXD101
Drug: Carfilzomib — Given intralesionally
  Other Names: Kyprolis; PR-171
Drug: Copanlisib Hydrochloride — Given intralesionally
  Other Names: 5-Pyrimidinecarboxamide, 2-Amino-N-(2,3-dihydro-7-methoxy-8-(3-(4-morpholinyl)propoxy)imidazo(1,2-C)quinazolin-5-yl)-, Hydrochloride (1:2); Aliqopa; BAY 80-6946 Dihydrochloride; BAY-80-6946 Dihydrochloride; Copanlisib Dihydrochloride
Biological: Daratumumab — Given intralesionally
  Other Names: Anti-CD38 Monoclonal Antibody; Darzalex; HuMax-CD38; JNJ-54767414
Drug: Fludeoxyglucose F-18 — Undergo FDG-PET
  Other Names: 18FDG; FDG; Fludeoxyglucose (18F); fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Drug: Gemcitabine Hydrochloride — Given intralesionally
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; FF 10832; FF-10832; FF10832; Gemcitabine HCI; Gemzar; LY-188011; LY188011
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Nivolumab — Given intralesionally
  Other Names: BMS-936558; CMAB819; MDX-1106; NIVO; Nivolumab Biosimilar CMAB819; ONO-4538; Opdivo
Biological: Obinutuzumab — Given intralesionally
  Other Names: Anti-CD20 Monoclonal Antibody R7159; GA-101; GA101; Gazyva; huMAB(CD20); R7159; RO 5072759; RO-5072759; RO5072759
Biological: Pembrolizumab — Given intralesionally
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Procedure: Positron Emission Tomography — Undergo FDG-PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging
Biological: Rituximab — Given intralesionally
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab ABBS; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; rituximab-abbs; RTXM83; Truxima
Drug: Romidepsin — Given intralesionally
  Other Names: Antibiotic FR 901228; Depsipeptide; FK228; FR901228; Istodax; N-[(3S,4E)-3-Hydroxy-7-mercapto-1-oxo-4-heptenyl]-D-valyl-D-cysteinyl-(2Z)-2-amino-2-butenoyl-L-valine, (4->1) Lactone, Cyclic
Other: Saline — Given intralesionally
  Other Names: ISOTONIC SODIUM CHLORIDE SOLUTION; Sodium Chloride 0.9%
Biological: Trastuzumab — Given intralesionally
  Other Names: ABP 980; ALT02; Anti-c-ERB-2; Anti-c-erbB2 Monoclonal Antibody; Anti-ERB-2; Anti-erbB-2; Anti-erbB2 Monoclonal Antibody; Anti-HER2/c-erbB2 Monoclonal Antibody; Anti-p185-HER2; c-erb-2 Monoclonal Antibody; HER2 Monoclonal Antibody; Herceptin; Herceptin Biosimilar PF-05280014; Herceptin Trastuzumab Biosimilar PF-05280014; Herzuma; Kanjinti; MoAb HER2; Monoclonal Antibody c-erb-2; Monoclonal Antibody HER2; Ogivri; Ontruzant; PF-05280014; rhuMAb HER2; RO0452317; SB3; Trastuzumab Biosimilar ABP 980; Trastuzumab Biosimilar ALT02; trastuzumab biosimilar EG12014; Trastuzumab Biosimilar HLX02; Trastuzumab Biosimilar PF-05280014; Trastuzumab Biosimilar SB3; Trastuzumab Biosimilar SIBP-01; Trastuzumab-anns; Trastuzumab-dkst; Trastuzumab-dttb; Trastuzumab-pkrb; Trastuzumab-qyyp; Trazimera

SUMMARY:
This pilot phase I trial studies the side effects of direct tumor microinjection and fludeoxyglucose F-18 positron emission tomography (FDG-PET) in testing drug sensitivity in patients with non-Hodgkin lymphoma, Hodgkin lymphoma, or stage IV breast cancer that has returned after a period of improvement or does not respond to treatment. Injecting tiny amounts of anti-cancer drugs directly into tumors on the skin or in lymph nodes and diagnostic procedures, such as FDG-PET, may help to show which drugs work better in treating patients with non-Hodgkin lymphoma, Hodgkin lymphoma, or breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the safety of in vivo in host drug sensitivity testing in patients with breast cancer and patients with lymphoma (nodal, extranodal masses, or cutaneous lesions).

SECONDARY OBJECTIVES:

I. To assess the feasibility of in vivo in host drug sensitivity testing in this patient population.

II. To identify targeted therapies with potential activity in relapsed lymphoma and metastatic breast cancer.

III. To evaluate the adverse event profile within each patient population.

CORRELATIVE OBJECTIVES:

I. To assess for apoptosis in response to intratumoral injection using known biomarkers (e.g., by morphology, Ki-67, caspace-3 assay as a marker of early apoptosis).

II. To evaluate intratumoral biomarkers, intratumoral cell populations, and distribution, identify potential biomarkers that correlate with response to therapy based on individual therapies.

OUTLINE:

Patients undergo FDG-PET and receive saline intralesionally on day 1. Patients also receive up to five additional injections of gemcitabine hydrochloride, romidepsin, belinostat, carfilzomib, copanlisib hydrochloride, nivolumab, trastuzumab, daratumumab, obinutuzumab, pembrolizumab, or rituximab intralesionally per investigator on day 1. Beginning 5 days later, patients with nodal/extranodal mass undergo restaging FDG-PET and biopsy (if clinically feasible). Within 3-7 days, patients with cutaneous disease undergo restaging photography and biopsy.

After completion of study treatment, patients are followed up at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Histologically proven of relapsed or refractory

  * Non-Hodgkin lymphoma (NHL) or Hodgkin lymphoma (HL) nodal or extranodal mass OR
  * Cutaneous T-cell lymphoma (CTCL) including mycosis fungoides (MF), as well as transformed MF OR
  * Breast adenocarcinoma with nodal or cutaneous metastases (stage 4)

    * NOTE: Patients must be refractory to or intolerant of existing therapy(ies) known to provide clinical benefit for their condition
    * NOTE: The patient must not be a candidate for any curative therapy or any known life-prolonging therapy
* Cohort I: For nodal/extranodal mass, presence of lesions that are amenable for injections as determined by interventional radiology

  * NOTE: Nodal or extranodal mass must be palpable and easily accessible; masses such as mediastinum, retroperitoneum, within solid organs, spinal sites, central nervous system (CNS) sites, etc., are NOT allowed
* Measurable disease:

  * For nodal or extranodal disease (lymphoma or breast): must have at least 2 lesions that are >= 20 mm (2.0 cm) in the longest diameter by physical exam and/or on cross-sectional imaging and measurable in two perpendicular dimensions per computed tomography PET-computed tomography (CT); For Cohort I, the lesions must be amenable to intralesional injections as determined by interventional radiology (including tumors that can be safely accessed using imaging guidance and treated with minimal risk to adjacent structures)
  * For cutaneous lesions (lymphoma or breast): at least two visible, non-infected skin lesions that are greater than 1 cm and are amenable to intralesional injection as determined by investigator
* Candidate for further therapy and able to wait 7 days prior to start of next systemic therapy
* Absolute neutrophil count (ANC) >= 1000/mm^3 (obtained =< 14 days prior to registration)
* Platelet count >= 50,000/mm^3 (obtained =< 14 days prior to registration)
* International normalized ratio (INR)/prothrombin time (PT) =< 1.5 (obtained =< 14 days prior to registration)
* Negative serum or urine pregnancy test done =< 7 days prior to registration, for persons of childbearing potential only
* Provide written informed consent
* Willing to return to enrolling institution for follow-up
* Willing to provide tissue samples for correlative research purposes

Exclusion Criteria:

* Any of the following:

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential who are unwilling to employ adequate contraception
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Systemic corticosteroids between pre-PET and post-PET evaluation and biopsy
* Prohibited treatments and or therapies

  * Autologous stem cell transplant (ASCT) =< 12 weeks prior to registration
  * Prior chemotherapy =< 2 weeks prior to registration
  * Prior treatment with nitrosureas =< 4 weeks prior to registration
  * Therapeutic anticancer antibodies =< 2 weeks prior to registration
  * Radio- or toxin immunoconjugates =< 4 weeks prior to registration
  * Radiation therapy to the injected area =< 2 weeks prior to registration
  * Major surgery =< 2 weeks prior to registration
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Requires anticoagulation that cannot be discontinued prior to biopsy

  * Note: Exception if able to hold antiplatelet agents 7 days prior to the injections and biopsy
  * NOTE: Low molecular weight heparin (LMWH) will be allowed for bridging if on warfarin
  * NOTE: Heparin for line patency without detectable lab abnormalities for coagulation will be allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2022-10-03 (Actual)

PRIMARY OUTCOMES:
Incidence of drug sensitivity as measured by injection site skin reaction | Up to 3 months
  Skin reactions will be assessed using the Cancer Therapy Evaluation Program (CTEP) active version of the Common Terminology Criteria for Adverse Events (CTCAE) and will consist of any grade 3 or higher treatment-related pain, skin or subcutaneous tissue disorders. Incidence rates of skin reactions will be estimated by the number of patients with reactions divided by the total number of evaluable patients per disease type. Exact binomial 95% confidence intervals for the true incidence rate will be calculated.

SECONDARY OUTCOMES:
Feasibility | Up to 3 months
  For Cohort I (Arms A & B) and Cohort II (Arm D): The study will be determined to be feasible if at least 70% of the enrolled patients complete the injection and response evaluation. The feasibility rate will be estimated by the number of patients completed divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true feasibility rate will be calculated. For Cohort II (Arm C): The feasibility rate will be evaluated for the device regarding whether the device will be able to target the affected lymph nodes in at least 50% of the time. The feasibility rate will be estimated by the number of patients completed divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true feasibility rate will be calculated.
Nodal disease response rate | Up to 5 days post injection
  Defined as a decrease in standardized uptake value (SUV) uptake by 25% at site of injection. Will be estimated by the number of injection sites with responses divided by the total number of injected sites. Exact binomial 95% confidence intervals for the true overall response rate will be calculated.
Cutaneous response rate based upon the modified Severity Weighted Assessment Tool score | Up to 7 days post injection
  Will be estimated by the number of injection sites with responses divided by the total number of injected sites. Exact binomial 95% confidence intervals for the true overall response rate will be calculated.
Incidence of adverse events | Up to 3 months
  Will be evaluated using the CTEP active version of the CTCAE. The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns.

OTHER OUTCOMES:
Apoptosis in response to intratumoral injection | Up to 3 months
  Will assess using morphology (evidence of necrosis), measurement by immunohistochemistry of Ki67 (a marker of cell proliferation) and cleaved Caspace-3.

CONTACTS AND LOCATIONS:
Overall Officials: Grzegorz S. Nowakowski, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials